CLINICAL TRIAL: NCT03114696
Title: Double-blind, Placebo-controlled, Randomised Pilot Clinical Trial to Explore Benefit and Tolerability of IQP-AO-101 in Healthy Subjects With Sleep Complaints
Brief Title: Benefit of IQP-AO-101 for Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INQ/020316
Record Dates: First submitted 2017-04-06; First posted 2017-04-14 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Insomnia, Nonorganic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IQP-AO-101 (Experimental): 1 dose (sachet) to be consumed 30 - 60 mins before bedtime
  Interventions: Dietary Supplement: IQP-AO-101
- Placebo (Placebo Comparator): 1 dose (sachet) to be consumed 30 - 60 mins before bedtime
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-AO-101 — 1 dose (sachet) to be consumed 30 - 60 mins before bedtime
  Arms: IQP-AO-101
Dietary Supplement: Placebo — 1 dose to be consumed 30 - 60 mins before bedtime. (Identical to investigational product)
  Arms: Placebo

SUMMARY:
The objective of this pilot clinical trial is to evaluate the potential of IQP-AO-101 with respect to sleep-promoting effects in subjects with sleep complaints.

ELIGIBILITY:
Inclusion Criteria:

1. 21-65 years old
2. Non-organic moderate sleep complaints in the last year prior to V1, as per investigator's judgement
3. Pittsburgh Sleep Quality Index (PSQI) score 6-15 at V1
4. Body mass index (BMI) 18.5-29.9 kg/m2
5. Generally in good health without clinically significant findings at V1
6. Readiness to comply with study procedures, in particular:

   * Consumption of the IP during the treatment period
   * Wearing activity tracker during the scheduled time periods
   * Filling in the subject diary
   * Keeping habitual diet and level of physical exercise, as well as smoking habits if applicable
7. Women of child-bearing potential:

   * Negative pregnancy testing (ß-HCG in urine) at V1
   * Commitment to use reliable contraception methods during the entire study
8. Written informed consent form

Exclusion Criteria:

1. Known sensitivity to any components of the investigational product
2. Insomnia (according to investigator's judgement))
3. Substantial daily sleepiness as per investigator's judgement
4. Less than 5 hours sleep per night on average, self-reported at V1
5. Any medical condition associated with sleep disorder as per investigator's judgement (e.g. sleep apnoea, restless legs syndrome, neurological / psychiatric disorder)
6. Any lifestyle and other factors potentially associated with sleep problems as per investigator's judgement (e.g. excessive caffeine intake, shift work, long-distance travelling, significant stressors such as active grieving etc.)
7. History and/or presence of clinically significant dis-ease, which per investigator's judgement could interfere with the results of the study or the safety of the subject:

   * Eating disorders such as anorexia
   * Untreated or non-stabilised metabolic diseases, e.g. diabetes mellitus
   * Untreated or non-stabilised thyroid disorder
   * Untreated or non-stabilised hypertension (regular systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg)
   * Significant gastrointestinal diseases
   * Any other known significant or serious condition / disease that renders subjects ineligible (e.g. history of malignancy within the past 5 years prior to V1, any clinically significant cardiovascular, renal, liver disease etc.)
8. Use of drugs/supplements which could interfere with the results of the study as per investigator's judgement (e.g. melatonin and melatonin derivatives, stimulants, neuroleptics, benzodiazepines, antidepressants, hypnotics) within the last 4 weeks prior to V1 and during the study
9. Behavioural intervention for sleep difficulties in the past 6 months and during the study as per investigator's judgement
10. Deviation of laboratory parameter(s) at V1 that is:

    * clinically significant or
    * >2x ULN (upper limit of normal), unless the deviation is justified by a previously known not clinically relevant condition, e.g. Gilbert's syndrome)
11. Alcohol abuse (men: ≥21 units/week, women: ≥14 units/ week; 1 unit equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
12. Drug abuse
13. Participation in another study during the last 4 weeks prior to V1 and during the study
14. Women of child-bearing potential: pregnant or breast-feeding
15. Any other reason for exclusion as per investigator's judgment, e.g. insufficient compliance with study procedures

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Change in mAIS parameters at V5 vs V2 | 6 weeks
  Change in modified Athens Insomnia Scale parameters

SECONDARY OUTCOMES:
Change in mAIS parameter at V3 and V4, vs V2 | 1 week, 4 weeks
  Change in modified Athens Insomnia Scale parameters
Change in activity tracker sleep parameters | 1 week, 6 weeks
  Use of an activity tracker to monitor sleep and compare against baseline
Change in FAIR-2 | 1 week, 4 weeks, 6 weeks
  Change in FAIR-2 at each visit

OTHER OUTCOMES:
Safety parameters assessed by number of subjects with abnormal laboratory values | 1 week, 4 weeks, 6 weeks
  Number of subjects with abnormal laboratory values
Adverse events that are related to treatment | 6 weeks
  Monitoring of adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Analyze & Realize, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bongartz U, Tan BK, Seibt S, Bothe G, Uebelhack R, Chong PW, Wszelaki N. Sleep Promoting Effects of IQP-AO-101: A Double-Blind, Randomized, Placebo-Controlled Exploratory Trial. Evid Based Complement Alternat Med. 2019 May 2;2019:9178218. doi: 10.1155/2019/9178218. eCollection 2019. PMID 31186669